CLINICAL TRIAL: NCT06631859
Title: The Effect of Cosmetic Products Containing Assam Tea (Camellia Sinensis Var. Assamica) Extracts on Irritation, Moisturization, Skin Elasticity, Wrinkles, and Satisfaction in Volunteers.
Brief Title: The Safety and Efficacy Assessment of Cosmetic Products Containing Assam Tea Extracts in Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 23258-17
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volunteers who recieved tested product (Experimental): Volunteers who recieved tested product
  Interventions: Other: Cosmetic products containing 2.5% Assam tea
- Volunteers who recieved base product (Placebo Comparator): Volunteers who recieved base product
  Interventions: Other: Cosmetic products containing 0% Assam tea

INTERVENTIONS:
Other: Cosmetic products containing 0% Assam tea — Cosmetic products containing 0% Assam tea
  Arms: Volunteers who recieved base product
Other: Cosmetic products containing 2.5% Assam tea — Cosmetic products containing 2.5% Assam tea
  Arms: Volunteers who recieved tested product

SUMMARY:
Thailand has entered an aging society, prompting increased research on improving the elderly quality of life and preventing age-related diseases, with a particular focus on skin aging. Skin aging is linked to the degradation of dermal and epidermal tissue, leading to decreased collagen, elastin, and glycosaminoglycans, which causes reduced skin elasticity and wrinkles.

Assam tea is native to northern Thailand and is traditionally used in local products like fermented "Miang." Research shows that Assam tea contains high levels of polyphenols, particularly catechins, which have strong antioxidant properties that help combat conditions such as cancer, cardiovascular disease, and skin aging.

The study aims to study the effect of cosmetic products from Assam tea on irritation, moisturization, skin elasticity, wrinkles, and satisfaction in volunteers to enhance its value, particularly for the elderly. This effort is intended to boost the local economy, promote community-based tourism, and expand Assam tea products to national and international markets, ultimately improving livelihoods and addressing environmental concerns in northern Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 years and older
* Good physical and mental health
* Willing and able to provide informed consent to participate and complete the entire duration of the study

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Presence of existing dermatological conditions
* History of autoimmune disorders
* Prior use of products related to wrinkle reduction or those containing active ingredients that stimulate collagen or elastin production, including topical and oral products used within the past three months (e.g., coenzyme Q10, marine extracts, pine bark extract, glutathione, and vitamin C)
* Participation in any other volunteer study or program within the past three months
* Use of the following medications within the past three months: contraceptives, phenytoin, hydantoin, levodopa, chloroquine, cancer chemotherapy drugs, or medications containing heavy metals
* History of receiving dermatological or cosmetic procedures such as IPL (Intense Pulse Light) laser, phonophoresis, iontophoresis, laser treatments, Botox injections, fillers, or stem cell injections
* Volunteers who exhibit sensitivity or irritation to the test products used in the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-03-17 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Skin hydration | 2 months
  Measure skin hydration by using a Corneometer®
Transepidermal water loss (TEWL) | 2 months
  Measure TEWL by using a Tewameter®
Skin irritation | 2 months
  Evaluate redness and edema occurred after applying the tested products by closed patch test under occlusion with Finn chamber®
Values from Cutometer® | 2 months
  Such as R0, R1, R2, R3, R4, R5, R6, R7, R8, R9
Values from Skin-Visiometer® | 2 months
  Such as Volume, Surface, SEr, SEsc, SEsm, SEw
Sensory evaluation | 2 months
  Measure the parameters such as color, odor, viscosity, texture, etc using labeled affective magnitude scale

CONTACTS AND LOCATIONS:
Locations (1):
- School of Cosmetic Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand